CLINICAL TRIAL: NCT06342154
Title: Does Endorphin Massage Applied Before Cesarean Section Reduce the Anxiety of Pregnant Women?
Brief Title: Does Endorphin Massage Reduce the Anxiety of Pregnant Women?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Yonca Çiçek Okuyan, Research Assistant, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCBU-SBF-YC-03
Record Dates: First submitted 2024-03-22; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related
Keywords: endorphin massage; cortisol level; stress; pregnant women

STUDY DESIGN:
Intervention Model Description: randomized study with experimental and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endorphin massage group (Experimental): The researcher will show husbands how to give endorphin massage to their pregnant wives. Additionally, they will be asked to choose one of three different instrumental relaxation music pieces played without lyrics to help them relax, and the chosen music will be sent to the pregnant women via WhatsApp. They will be instructed to play the music while performing the endorphin massage. Husbands of pregnant women in the experimental group will be asked to apply a total of 20 minutes of endorphin massage within 1 hour, divided into two sessions of 10 minutes each.
  Interventions: Behavioral: Endorphin Massage
- routine care group (No Intervention): They will receive routine nursing care.

INTERVENTIONS:
Behavioral: Endorphin Massage — The person who will perform the endorphin massage opens his hands with his palms facing himself and draws a semicircle with the nails of his middle, ring and little fingers touching the sacrum. Then, a semicircle is drawn with the fingertips from each side of the spine, starting from the sacrum to the shoulder area, towards the waist area, As a result of this process, a palm shape is drawn on the back. Effleurage is applied from the shoulders to the arms up to the elbows. Effleurage is applied towards the shoulders by pressing from the elbows upwards with the back of the thumb. Effleurage is applied up to the sacrum by pressing circular movements with two thumbs on both sides of the spine. Effleurage is applied from the sacrum to the neck by pressing with two thumbs in a circular motion on both sides of the spine (approximately 1.5 cm apart). Lastly, effleurage is applied to the neck area and scalp, then petrissage (rubbing) is applied and the massage is completed.
  Arms: endorphin massage group

SUMMARY:
Before cesarean section surgery, researchers will demonstrate endorphin massage to the husbands of pregnant women, and they will be asked to apply the massage before the surgery. The stress levels and pain levels of women will be compared before and after the massage.

DETAILED DESCRIPTION:
The sample size of the research was calculated using G*Power 3.1.9.4 software as a minimum of 34 with 95% power, 0.01 alpha, and 0.9 effect size. The sample size was planned as experimental (n=34) and control (n=34) groups. To ensure the equality of the samples in both groups, a simple randomization method was used, where pregnant women with odd hospital protocol numbers will be included in the experimental group and those with even numbers will be included in the control group. Pregnant women who are admitted for pre-cesarean section care will be informed about the study, and their voluntary consent will be obtained both in written and verbal form. Pre-tests will be administered to both the experimental and control groups at 08:00, and blood samples will be taken to measure cortisol levels. Subsequently, an intervention will be applied to those in the experimental group, while those in the control group will receive routine nursing care. At 09:00, post-tests will be administered to both the experimental and control groups, and blood samples will be taken again to measure cortisol levels. The pre-test and post-test results, as well as the mean cortisol levels, will be compared between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Being admitted to the hospital for cesarean section
* Being willing to participate in the research

Exclusion Criteria:

* Having psychiatric illness
* native language not Turkish

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 68 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-10-09 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) | one hour after intervention
  VAS is preferred to convert some values that cannot be measured numerically into numerical values. VAS, which is a simple, effective, repeatable pain intensity measurement method that requires minimal tools, provides rapid measurement of pain intensity under clinical and laboratory conditions. There are studies in which VAS is used to evaluate pain in prenatal patients. In VAS, the patient is asked to make a mark on a 10 cm horizontal line that shows his current situation. In this study, for pain; Markings are made on a 10 cm horizontal line, one end of which indicates that the patient's pain is very good (0 = no pain), and the other end indicates that the patient's pain is very bad (10 = the most severe). The length of the distance from the point where there is no pain (0) to the point marked by the patient shows the patient's pain intensity.
State and Trait Anxiety Scales | one hour after intervention
  It is used to determine state and trait anxiety levels in individuals. State-Trait Anxiety Scale consists of a total of 40 items, 20 items each. The State Anxiety Scale requires the individual to describe how he or she feels at a particular moment and under certain circumstances. The total score of the scale varies between 20-80. A high score from the scale indicates a high level of anxiety, and a low score indicates a low level of anxiety.
cortisol level | one hour after intervention
  A high cortisol level indicates high stress, while a low level indicates low stress. Since cortisol levels follow a circadian rhythm, the timing of evaluation is crucial. Therefore, the first assessment in the study was conducted at 08:00, and the final evaluation was performed at 09:00.

CONTACTS AND LOCATIONS:
Overall Officials: Yonca Çicek, PhD, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar Üniversitesi Hafsa Sultan Hastanesi, Manisa, Turkey (Türkiye)